CLINICAL TRIAL: NCT05968612
Title: A Single-Dose, Bioequivalence and Food Effect Bioavailability Study in Healthy Volunteers Comparing the Commercial Lumacaftor 200 mg / Ivacaftor 125 mg Combination Film-Coated Tablet (Orkambi®) to the Lumacaftor 200 mg Film-Coated Tablet Formulation, and the Lumacaftor 200 mg Film-Coated Tablet Formulation in the Fasted to Fed State.
Brief Title: Bioequivalence and Food Effect Bioavailability Study of Lumacaftor Film-Coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qanatpharma Canada LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: QP586-01
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteer
Keywords: lumacaftor; cystic fibrosis transmembrane regulator-corrector; CFTR-corrector; food effect; healthy volunteers; cerebral blood flow; CBF
MeSH Terms: interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Treatment A (Test-Fed) (Experimental): Following a 10-hour overnight fasting period, subjects will eat a high-fat, high-calorie breakfast, and 30 minutes later subjects will receive a single dose of 2 Lumacaftor 200 mg Film-Coated Tablets.
  Interventions: Drug: Lumacaftor 200 mg Film-Coated Tablet Formulation
- Treatment B (Reference-Fed) (Active Comparator): Following a 10-hour overnight fasting period, subjects will eat a high-fat, high-calorie breakfast, and 30 minutes later subjects will receive a single dose of 2 Lumacaftor 200 mg/Ivacaftor 125 mg Combination Film-Coated Tablets (Orkambi®)
  Interventions: Drug: Lumacaftor 200 mg/Ivacaftor 125 mg Film-Coated Tablet
- Treatment C (Test-Fasted) (Experimental): Following a 10-hour overnight fasting period, subjects will receive a single dose of 2 Lumacaftor 200 mg Film-Coated Tablets.
  Interventions: Drug: Lumacaftor 200 mg Film-Coated Tablet Formulation

INTERVENTIONS:
Drug: Lumacaftor 200 mg/Ivacaftor 125 mg Film-Coated Tablet — Film-coated tablet administered orally.
  Arms: Treatment B (Reference-Fed)
Drug: Lumacaftor 200 mg Film-Coated Tablet Formulation — Film-coated tablet administered orally.
  Arms: Treatment A (Test-Fed); Treatment C (Test-Fasted)

SUMMARY:
The objective of this study is to assess bioequivalence of lumacaftor from Lumacaftor 200 mg Film-Coated Tablet Formulation (Qanatpharma) versus the reference commercial product, Lumacaftor 200 mg /Ivacaftor 125 mg Combination Film-Coated Tablet (Orkambi®) in the fed state, and food-effect bioavailability of Lumacaftor 200 mg Film-Coated Tablet Formulation (Qanatpharma) in the fasted and fed state in healthy, non-smoking, male and non-pregnant female volunteers, 18 to 55 years of age, inclusive.

DETAILED DESCRIPTION:
This single-dose, randomized, open-label, three-way crossover, three-period, three-sequence, three-treatment, single-centre, bioequivalence and food-effect study will compare lumacaftor from Lumacaftor 200 mg Film-Coated Tablet test formulation and the commercial product, Lumacaftor 200 mg/Ivacaftor 125 mg Combination Film-Coated Tablet (Orkambi®) under fed conditions, and food-effect bioavailability study of Lumacaftor 200 mg Film-Coated Tablet test formulation from fasted to fed state.

The products will be studied using a crossover design with 39 healthy, non-smoking male and non-pregnant female volunteers being administered an oral dose of 1 x (2 x lumacaftor 200 mg) under fasted and fed conditions and 1 x (2 x lumacaftor 200 mg/ ivacaftor 125 mg) under fed conditions. There will be at least a 14-day washout period between the study periods to avoid carry-over effects of the preceding treatments.

This study is being conducted to support development of a lumacaftor mono-substance treatment for improving cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking male and non-pregnant female volunteers, 18 years to 55 years of age, inclusive.
2. Body mass index (BMI) that is between 18.5 and 30.0 kg/m^2, inclusive.
3. Results of clinical laboratory tests are within the normal range or with a deviation that is not considered clinically significant by the principal investigator.
4. Ability to fast for at least 10 hours and consume a high-fat, high-calorie meal, as well as standard meals.
5. Agree not to have a tattoo or body piercing until the end of the study.
6. Agree not to receive the COVID-19 vaccination from 7 days prior to the first study drug dose until 7 days after the last study drug administration in the study.
7. Female subjects of childbearing potential and males who are able to father children must meet the criteria defined in the protocol.

Exclusion Criteria:

1. Known history or presence of any clinically significant diseases or conditions unless determined as not clinically significant by the Investigator.
2. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the Investigator.
3. Presence of any significant physical or organ abnormality as determined by the Investigator.
4. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol breath test and cotinine. Positive pregnancy test for female subjects.
5. Known history or presence of:

   * Alcohol abuse or dependence within one year prior to first drug administration;
   * Drug abuse or dependence;
   * Hypersensitivity or idiosyncratic reaction to lumacaftor and ivacaftor, its excipients, and/or related substances;
   * Food allergies
   * Presence of any dietary restrictions unless deemed by the Investigator as "Not Clinically Significant".
   * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
6. Intolerance to and/or difficulty with blood sampling through venipuncture.
7. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets, etc.
8. Individuals who have donated, in the days prior to first study drug administration:

   * 50-499 mL of blood in the previous 30 days;
   * 500 mL or more in the previous 56 days.
9. Donation of plasma by plasmapheresis within 7 days prior to first study drug administration.
10. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.
11. Females having used implanted, injected, intravaginal, or intrauterine hormonal contraceptive within 6 months prior to first study drug administration.
12. Females taking oral or transdermal hormonal contraceptives within 30 days prior to first study drug administration.
13. Use of any enzyme-modifying drugs or products in the previous 30 days before first study drug administration.
14. Use of any prescription medication within 14 days prior to first study drug administration (except medically acceptable contraceptive products).
15. Use of any over-the-counter medications within 14 days prior to first study drug administration (except for medically acceptable contraceptive products).
16. Consumption of food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.
17. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing.
18. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by Investigator.
19. Difficulty with swallowing whole film-coated tablet.
20. Women who are pregnant or lactating.
21. Have had a tattoo or body piercing within 30 days prior to first study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
The maximal observed plasma concentration (Cmax) | Up to 72 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected pre-dose at 0, and post-dose at 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24, 48, and 72 hours
Area under the concentration-time curve from time zero to 72 hours (AUC72) | Up to 72 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected pre-dose at 0, and post-dose at 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24, 48, and 72 hours
Area under the concentration-time curve from time zero to infinity (AUCinf) | Up to 72 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected pre-dose at 0, and post-dose at 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24, 48, and 72 hours
Time when the maximal plasma concentration is observed (Tmax) | Up to 72 hours post dose in each treatment period
  Serial blood samples for determination of study drug will be collected pre-dose at 0, and post-dose at 0.25, 0.5, 0.75, 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 24, 48, and 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Szeto, MD, CCFP, Principal Investigator — BioPharma Service Inc.
Locations (1):
- BioPharma Services Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qanatpharma will provide access upon request to individual de-identified participant data reported in the publication beginning 12 months after publication and for up to 36 months following article publication. Data sharing requests can be made by qualified researchers for approved proposals under the terms of a Data Use Agreement. Contact information will be provided at the time of article publication.
Supporting Information: Study Protocol
Time Frame: 12 months after article publication and for up to 36 months following article publication
Access Criteria: Data sharing requests can be made by qualified researchers for approved proposals under the terms of a Data Use Agreement.

REFERENCES:
- [Derived] Papaelias A, Lidington D, Bolz SS. Demonstrating Bioequivalence for a Lumacaftor Monosubstance Formulation Versus Orkambi(R) (Lumacaftor/Ivacaftor) in Healthy Subjects. Drugs R D. 2025 Sep;25(3):221-229. doi: 10.1007/s40268-025-00514-9. Epub 2025 Jun 23. PMID 40551045